CLINICAL TRIAL: NCT00291395
Title: PGI2 Induced Headache and Cerebral Haemodynamics in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: KA05055
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-09

CONDITIONS: Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders

INTERVENTIONS:
Drug: PGI2

SUMMARY:
Before , during and after intravenous administration of PGI2 we score/measure headache, rCBF, blood flow in middle cerebral artery and diameter of superficial temporal artery/radial artery and correlate that to known patophysiology of headache to see if PGI2 is involved in headache pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers,

Exclusion Criteria:

* Primary headache,
* headache on the day of investigation,
* Hypertension,
* hypotension,
* pregnant/nursing
* Daily intake of medication (except oral contraceptives)
* Cardiovascular or CNS disease
* Drug/Alcohol abuse
* Psychiatric disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-09

PRIMARY OUTCOMES:
Headache

SECONDARY OUTCOMES:
rCBF, blood flow, diameter of STA/RA, HR, BP

CONTACTS AND LOCATIONS:
Overall Officials: Troels Wienecke, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Glostrup, Denmark